CLINICAL TRIAL: NCT00720694
Title: Placebo Controlled Study to Investigate the Effectiveness and Safety of Extracorporeal Shock Wave Therapy in Unsuccessful Conservatively Treated Subject Suffering From Painful Heel Syndrome
Brief Title: Study of Effectiveness and Safety of Extracorporeal Shock Wave Therapy (ESWT) for Treatment of Painful Heel Syndrome
Acronym: ESWT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Storz Medical AG (Industry)
Responsible Party: Dr. Pavel Novak, Director Product Development, Storz Medical AG
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMS2005
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Verum (Active Comparator): Device: Duolith SD1 (Storz Medical AG) - Focused Extracorporeal shock wave therapy.
  The total energy flux density was increased continuously from 0.01 to 0.25 mJ/mm 2 within 500 introductory impulses. Thereafter, 2000 treatment impulses with 0.25 mJ/mm 2 (four impulses per second) were administered per session,and the interventionwas repeated up to a total of three sessions in weekly intervals.
  Interventions: Device: Duolith SD1
- Placebo / Sham (Sham Comparator): Sham Duolith SD1 (Storz Medical AG). The placebo group received identical sham intervention with an air- filled standoff that prevented the transmission of shock waves. The placebo handpiece was identical in design, shape, and weight to ensure that there was no way for the participants to identify the placebo handpiece.
  Interventions: Device: Sham Duolith SD1

INTERVENTIONS:
Device: Duolith SD1
  Other Names: Extracorporeal shock wave therapy; ESWT
  Arms: Verum
Device: Sham Duolith SD1
  Arms: Placebo / Sham

SUMMARY:
The purpose of this study is to determine if the Storz Duolith SD1 is more effective than placebo for treatment of heel pain syndrome for patients who have failed conservative treatment with other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* ability of subject or legal respondent to give written informed consent
* signed informed consent
* diagnosis of painful heel syndrome
* 6 months of unsuccessful conservative treatment
* washout from conservative treatment
* scores of 5 or greater on three VAS scales
* score of 3 or 4 on Roles and Maudsley Scale
* willingness to refrain from specified concomitant therapies
* willingness to keep subject diaries
* negative urine pregnancy test (if applicable) required use of contraception (if applicable)

Exclusion Criteria:

* tendon rupture, neurological or vascular insufficiencies
* inflammation of lower and upper ankle
* history of rheumatic disease, collagen, or metabolic disorders
* history of hyperthyroidism
* active malignant disease with or without metastasis
* Paget disease or calcaneal fat pad atrophy
* osteomyelitis
* fracture of calcaneus
* immunosuppressive therapy
* long term (6 months or greater) treatment with corticosteroid
* insulin dependent diabetes, severe cardiac or respiratory disease
* coagulation disorder or therapy with anticoagulants or antiplatelet drugs
* bilateral painful heel
* planned treatment within 8 weeks of enrollment that may confound pain results
* less than required washout of other treatments
* previous surgery for painful heel
* previous unsuccessful treatment for painful heel with shock wave device
* history of allergy or hypersensitivity to local anesthetics
* significant abnormalities of hepatic function
* poor physical condition
* pregnant female
* active infection or history of chronic infection in treatment area
* history of peripheral neuropathy
* history of systemic inflammatory disease
* history of worker's compensation or litigation
* participation in study of investigational device within 30 days of selection or current active study participation
* in the opinion of the investigator, inappropriate for study inclusion
* unwilling to comply with study requirements
* implanted pacemaker, insulin pump, defibrillator, or neurostimulator
* implanted prosthetic device in area of treatment
* open wounds or skin rashes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Heel pain composite score | Follow-Up 1
  Sum of three VAS scales
Roles and Maudsley Score | Follow-Up 1
  functional improvement on a four-level grading scale: excellent indicates no pain, full movement, and activity; good indicates occasional discomfort, full move- ment, and activity; fair indicates some discomfort after prolonged activity; and poor indicates pain-limiting activities.

SECONDARY OUTCOMES:
Physician judgement of effectiveness | Follow-Up 1
  5-point scale ranging from very good to poor
Subject satisfaction with treatment | Follow-Up 1
  7-point scale ranging from very satisfied to very unsatisfied
Rate of success | Follow-Up 1
  at least 60% pain reduction in the single VAS scores
Rate of success | Follow-Up 2
  at least 60% pain reduction in the single VAS scores
Overall rate of success with regard to heel pain | Follow-Up 1
  at least 60% decrease of heel pain in at least two of the three VAS measurements
Roles and Maudsley score rate of success | Follow-Up 1
  rating of excellent or good
consumption of concomitant analgesic medication | Follow-Up 1
  medication
Heel pain composite score | Follow-Up 2
  Sum of three VAS scales
Roles and Maudsley Score | Follow-Up 2
  functional improvement on a four-level grading scale: excellent indicates no pain, full movement, and activity; good indicates occasional discomfort, full move- ment, and activity; fair indicates some discomfort after prolonged activity; and poor indicates pain-limiting activities.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Palo Alto Medical Fondation, Palo Alto, California
  - Connecticut Orthopedics Specialists, Hamden, Connecticut
  - Advanced Footcare Specialists of Connecticut, LLC, Newtown, Connecticut
  - Galli Podiatric Foot and Ankle Associates, New York, New York
  - Ankle and Foot Care Centers, Boardman, Ohio
  - The Sports Medicine Clinic, Seattle, Washington

REFERENCES:
- [Result] Gollwitzer H, Saxena A, DiDomenico LA, Galli L, Bouche RT, Caminear DS, Fullem B, Vester JC, Horn C, Banke IJ, Burgkart R, Gerdesmeyer L. Clinically relevant effectiveness of focused extracorporeal shock wave therapy in the treatment of chronic plantar fasciitis: a randomized, controlled multicenter study. J Bone Joint Surg Am. 2015 May 6;97(9):701-8. doi: 10.2106/JBJS.M.01331. PMID 25948515